CLINICAL TRIAL: NCT01519401
Title: Clinical Efficacy and Metabolic Impact of Two Different Dosages of Ethinyl-estradiol in Association With Drospirenone in Normal-weight Women With Polycystic Ovary Syndrome: a Randomized Study.
Brief Title: Effect of Two Different Dosages of Ethinyl-estradiol in Association With Drospirenone in Women With Polycystic Ovary Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Maurizio Guido, medical doctor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000102010
Record Dates: First submitted 2012-01-23; First posted 2012-01-26 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Polycystic Ovary Syndrome; Estro-progestin Drugs
Keywords: PCOS; drospirenone ethinylestradiol; androgens; metabolism
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — drospirenone; Ethinyl Estradiol

ARMS (2):
- 3 mg drospirenone and 20 µg ethinyl-estradiol (Active Comparator)
  Interventions: Drug: 3 mg drospirenone and 20 µg ethinyl-estradiol
- 3 mg drospirenone and 30 µg ethinyl-estradiol (Active Comparator)
  Interventions: Drug: 3 mg drospirenone and 30 µg ethinyl-estradiol

INTERVENTIONS:
Drug: 3 mg drospirenone and 20 µg ethinyl-estradiol
  Arms: 3 mg drospirenone and 20 µg ethinyl-estradiol
Drug: 3 mg drospirenone and 30 µg ethinyl-estradiol
  Arms: 3 mg drospirenone and 30 µg ethinyl-estradiol

SUMMARY:
The estrogenic component of estro-progestin (EP) is responsible for a negative impact on the metabolic and lipid assessment in women with polycystic ovary syndrome (PCOS).

The objective of this study is to compare the effects of a long term administration of two EP combinations, containing the same progestin (3 mg drospirenone) and a different dose of ethinyl-estradiol (EE) (20 vs 30 μg ) on the clinical and endocrine-metabolic parameters in normal weight PCOS women. The investigators enrolled 30 patients, randomly allocated to group A (20 µg EE - 3 mg DRSP) and 15 to group B (30 µg EE - 3 mg DRSP). Hirsutism score evaluation, hormonal assays, oral glucose tolerance test, euglycaemic hyperinsulinaemic clamp and lipid profile were performed at baseline and after 6 and 12 months of therapy.

ELIGIBILITY:
Inclusion Criteria:

* normal weight women with Polycystic ovary syndrome, diagnosed in accordance with Rotterdam Consensus Conference Criteria 2003.

Exclusion Criteria:

* pregnancy
* past history of cardiovascular disease, diabetes mellitus (or impaired glucose tolerance as determined by a standard 75 g oral glucose tolerance test), hypertension
* significant liver or renal impairment
* other hormonal dysfunction (hypothalamic, pituitary, thyroidal or adrenal causes for the clinical signs)
* neoplasms
* unstable mental illness

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To compare the effects of two EP combinations on endocrine-metabolic parameters in normal weight PCOS women | twelve months
  hormonal assays, oral glucose tolerance test, euglycaemic hyperinsulinaemic clamp and lipid profile

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Sacred Heart, Rome, Italy

REFERENCES:
- [Derived] Romualdi D, De Cicco S, Busacca M, Gagliano D, Lanzone A, Guido M. Clinical efficacy and metabolic impact of two different dosages of ethinyl-estradiol in association with drospirenone in normal-weight women with polycystic ovary syndrome: a randomized study. J Endocrinol Invest. 2013 Sep;36(8):636-41. doi: 10.1007/BF03346756. PMID 24105072